CLINICAL TRIAL: NCT00966303
Title: The Effectiveness of a Cardiac Rehabilitation in Patients With Cardiomyopathy
Brief Title: Cardiac Rehabilitation in Cardiomyopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fortaleza University (Other)
Collaborators: Edson Queiroz Foundation (Unknown)
Responsible Party: Davi Simões Sales, Fortaleza University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FR150091
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Cardiomyopathies
Keywords: rehabilitation; dyspnea; strength
MeSH Terms: conditions — Cardiomyopathies; Dyspnea | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cardiac Rehabilitation (Experimental): 9 patients with cardiomyopathy in functional class III or IV, submitted to an 8-week program with exercises and respiratory muscle training.
  Interventions: Other: Cardiac Rehabilitation with diaphragmatic muscle training

INTERVENTIONS:
Other: Cardiac Rehabilitation with diaphragmatic muscle training — Stretching and aerobic exercises and respiratory muscle training with a Threshold ® device, with load of 40% of the maximal inspiratory pressure (MIP), two times a week during one hour.

SUMMARY:
This quantitative study aimed to evaluate the respiratory muscle strength, pulmonary function, cardiovascular function, and impact on quality of life in patients after cardiac rehabilitation associated with the diaphragmatic muscle training.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cardiomyopathies in functional class III or IV (New York Heart Association)
* Aged over 18 years
* Body mass index below 30 kg/m2

Exclusion Criteria:

* Confused and depressed patients
* Cardiac instability and worsening dyspnea after initiation of treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The effectiveness of a cardiac rehabilitation in patients with cardiomyopathy, evaluating the respiratory muscle strength, pulmonary function, cardiovascular function, and impact on quality of life. | 8 weeks / Twice a week

CONTACTS AND LOCATIONS:
Overall Officials: Davi S Sales, Bachelor, Principal Investigator — Fortaleza University; Daniela GB Mont'Alverne, Doctor, Study Director — Fortaleza University
Locations (1):
- Fortaleza University - Nucleus of Integrated Medical Attention, Fortaleza, Ceará, Brazil